CLINICAL TRIAL: NCT03751865
Title: Early Detection and Intervention for Women At-risk of Psychosis in Hong Kong: A Randomized Controlled Trial
Brief Title: Early Detection and Intervention for Women At-risk of Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Eric Y.H. Chen, Chi-li Pao Foundation Professor of Psychiatry; Chair Professor in Psychiatry; Head, Department of Psychiatry, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JCWowCBT; UW 18-231 (Other: HKU/HKW IRB)
Record Dates: First submitted 2018-06-14; First posted 2018-11-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Prodromal Schizophrenia
MeSH Terms: conditions — Schizotypal Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT group (Experimental): This intervention aims for distress reduction, symptom coping, and life quality enhancement. It is a gender-specific CBT tailor-made for the at-risk population. The intervention is delivered by a registered clinical psychologist.
  Interventions: Behavioral: CBT
- Psychoeducation group (Active Comparator): The content of the psycho-education program will be related to healthy living content and mental health knowledge, such as food hygiene, psychological well-being, knowledge about psychosis and common mental disorder and food nutrition. In addition, a weekly call to remind the subject about healthy living will also be provided to the subjects. The intervention is delivered by a registered social worker.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: CBT — A total of 8 CBT sessions will be provided to the participants, each session lasts for approximately 1.5 hour.
  Arms: CBT group
Behavioral: Psychoeducation — A total of 8 psychoeducation sessions will be provided to the participants, each session lasts for approximately 1.5 hour.
  Arms: Psychoeducation group

SUMMARY:
This study aims to examine the effectiveness of the cognitive behavioral therapy in preventing the conversion of psychosis in a sample of individuals at-risk for psychosis.

DETAILED DESCRIPTION:
Eligible subjects with informed consent provided will be randomly assigned to the cognitive behavioural therapy (CBT) group or psychoeducation group. Each group consists of 8 session spanning for 8 week.

ELIGIBILITY:
Inclusion Criteria:

* women of age 18-64
* at-risk mental state as defined by the Comprehensive Assessment of At-Risk Mental States (CAARMS)
* with an informed consent
* able to understand Cantonese and read/write Chinese

Exclusion Criteria:

* those mental conditions that requires other treatment priorities (e.g., suicidal risk, substance abuse, current or past episodes of psychotic disorder, personality disorders)
* those medical conditions that severely limits participation, comprehension, or adherence to the treatment (e.g., epilepsy, dementia, terminal medical illness);
* those who are receiving structured psychotherapy or counselling

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Functioning: Measured by Social and Occupational Functioning Assessment Scale (SOFAS) | Changes from baseline to immediate, 6- and 12-month post-intervention
  Measured by Social and Occupational Functioning Assessment Scale (SOFAS). The SOFAS is an observer rating scale. Ratings should be based on subject's behavior during the last 1 month. The score ranges from 0-100. A higher score represents a better outcome.
Functioning: Measured by Role Functioning Scale (RFS) | Changes from baseline to immediate, 6- and 12-month post-intervention
  Measured by Role Functioning Scale (RFS). The RFS is comprised of four single rating scaled for evaluating the functioning of individuals in specified areas of everyday life. The four role functions assessed are:(1)Working: productivity, (2) Independent living and self care, (3) Immediate social network relationships, and (4) Extended social network relationship. The values on each of the four scales range from 1 (minimal level of role functioning), to 7 (hypothetically optimal level of role functioning). Each of the seven points on the scales is accompanied by a behaviorally defined description.
Conversion of psychosis | 12-month post-intervention
  Proportion of subject that convert from at-risk state to psychosis

SECONDARY OUTCOMES:
Positive psychotic symptoms | Immediate, 6- and 12-month post-intervention
  Measurement of positive symptoms using the Chinese version of the Psychotic Symptom Rating Scales (C-PSYRATS). It comprises of the auditory hallucinations (AHS) and delusions subscales (DS). The AHS has 11 questions and the DS consists of 6 questions, each question has the responses ranging from 0-4. The higher score represents more severe positive psychotic symptoms.
Beliefs about the auditory hallucination | Immediate, 6- and 12-month post-intervention
  Measured by the Beliefs About Voices Questionnaire (BAVQ-R). The BAVQ-R has 35 questions, the 4 responses range from disagree, unsure, slightly agree to strongly agree. The higher score represents more convicted belief about the voices.
Depressive symptoms | Immediate, 6- and 12-month post-intervention
  Measured by the Calgary Depression Scale for Schizophrenia (CDSS). The scale consists of 9 questions, each has the response ranging from 0 to 3. The higher score presents more severe depressive symptoms.
Social anxiety :Measured by Liebowitz Social Anxiety Scale (LSAS) | Immediate, 6- and 12-month post-intervention
  Measured by Liebowitz Social Anxiety Scale (LSAS). The LSAS consists of 24 questions, the rater has to rate from 0-3 in Fear or Anxiety domain or Avoidance domain for each of the 24 questions. The higher score represents more severe social anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Yu Hai Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No